CLINICAL TRIAL: NCT03194139
Title: A Phase 1, Randomized, Double-Blind, Crossover, Single Dose Study Designed to Compare the Safety and Pharmacokinetics of Intravenously Administered Superoxide Dismutase Mimetic GC4711 and GC4419 in Healthy Volunteers
Brief Title: A Study Designed to Compare the Safety and Pharmacokinetics of Intravenously Administered Superoxide Dismutase Mimetic GC4711 and GC4419 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI-4711-001
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers; Healthy
Keywords: Healthy Adult; Superoxide Dismutase; First in Human; Free Radical Dismutase
MeSH Terms: interventions — avasopasem manganese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sentinel Cohort (Experimental)
  Interventions: Drug: GC4711 30 mg IV
- Crossover Design (Experimental)
  Interventions: Drug: GC4711 50 mg IV; Drug: GC4419 45 mg IV

INTERVENTIONS:
Drug: GC4711 30 mg IV — GC4711 will be infused IV as a single dose of 30 mg (3 mL GC4711 at 10 mg/mL) in 245 mL normal saline, totaling 250 mL, over a 60-minute period using a programmable pump
  Arms: Sentinel Cohort
Drug: GC4711 50 mg IV — GC4711 will be infused IV as a single dose of 50 mg (5 mL GC4711 at 10 mg/mL) in 245 mL normal saline, totalling 250 mL, over a 60-minute period using a programmable pump.
  Arms: Crossover Design
Drug: GC4419 45 mg IV — GC4419 will be infused IV as a single dose of 45 mg (5 mL GC4419 at 9 mg/mL) in 245 mL normal (0.9%) saline, totalling 250 mL, over a 60-minute period using a programmable pump.
  Arms: Crossover Design

SUMMARY:
The study will be a double-blind, randomized, crossover, single-dose assessment of IV-administered GC4711 compared to GC4419 in healthy volunteers.

Consenting subjects will undergo screening procedures within 28 days of the start of dosing. Pharmacokinetics (parent drug and major metabolites) will be assessed in plasma and urine from all subjects.

Initially, a sentinel cohort of 4 subjects, will be enrolled; each eligible subject will receive single dose of GC4711 IV at dose of 30 mg over one hour. Following a clinical safety review by the Galera study team , if no safety concerns are identified after the last subject completes study participation, enrollment will continue in 2 stages to a crossover study design. In stage 1, 12 subjects will be enrolled and in stage 2, if no safety concerns are identified in stage 1 following a clinical safety review by the Galera study team, 20 subjects will be enrolled. In both enrollment stages, eligible subjects in the crossover design will be randomized in 1:1 ratio to one of two treatment sequences: Test (GC4711) -> Ref (GC4419) or Ref (GC4419) -> Test (GC4711). On Day 1, subjects will receive the first treatment they were randomized to, and on Day 4 (following a washout), they will receive the second treatment. Subjects will be followed up for 2 days after the second treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18 and 50 years (inclusive) of age;
2. Subjects who provide written informed consent to participate in the study
3. Body Mass Index (BMI) 18 to 32 kg/m2 (inclusive) and weighing at least 50 kg during Screening and at Baseline.
4. Subjects in general good health
5. Chest X-ray free of clinically significant abnormalities
6. Blood pressure and heart rate within normal limits
7. Female subjects must:

   1. Have a negative pregnancy test during Screening and Baseline
   2. Be non-lactating
   3. Be at least two years postmenopausal, surgically sterile or practicing effective contraception

Exclusion Criteria:

1. History of clinically significant illness, disease, medical condition, or laboratory abnormality
2. Known hypersensitivity and/or allergy to study drugs
3. Use of any prescription or over-the-counter medication within one week prior to baseline;
4. Anticipated need for any medication during the course of the study
5. Use of nitrates or erectile dysfunction drugs such as phosphodiesterase type 5 (PDE 5) inhibitors (e.g., sildenafil, tadalafil, or similar agents), from 24 hours prior to screening throughout participation in the study;
6. Use of or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure, from 24 hours prior to screening throughout participation in the study;
7. Use of any vitamin or mineral supplement 24 hours prior to dosing, or anticipated use of any vitamin or mineral supplement throughout the duration of the study;
8. Positive HIV, Hepatitis B or Hepatitis C
9. Known history of substance abuse, drug addiction, or alcoholism within 3 years prior to Baseline;
10. Anticipated inability to abstain from alcohol, tobacco, or caffeine use from 48 hours prior to the administration of study drug and throughout the duration of the study;
11. History of smoking or any use of a tobacco product within six months prior to Baseline;
12. Donation of blood or blood products within 30 days prior to the Baseline;
13. Receipt of an investigational test substance within three months prior to the first dose of study drugs or anticipated receiving any study drugs (including placebo on another investigational study)
14. Subject has previously participated in this study, or in a prior study of GC4419 or GC4702.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-24 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Frequency, duration, and severity of adverse events (AEs) | From first dose of study medication until up to 3 days post last dose. Up to 6 days total
Incidence of clinically significant laboratory abnormalities | From first dose of study medication until up to 3 days post last dose. Up to 6 days total

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Holmlund, MD, Study Chair — Galera Therapeutics
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No